CLINICAL TRIAL: NCT04096261
Title: The Importance of Sleep Quality and the Blood-brain Barrier in Cognitive Disorders and Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: Resources had to be focused on other projects.
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Arda Can Cetindag (Unknown); Lukas Preis (Unknown)
Responsible Party: Principal Investigator, Oliver Peters, MD, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: BBB-Sleep
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Blood Brain Barrier Defect; Sleep Deprivation; Sleep Apnea; Alzheimer Disease
MeSH Terms: conditions — Sleep Deprivation; Sleep Apnea Syndromes; Alzheimer Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Cerebro-spinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy controls: Healthy controls recruited through public advertisement.
  Interventions: Diagnostic Test: Diagnostic Test
- Siblings of people with Alzheimer's dementia: Siblings of people with Alzheimer's dementia recruited through public advertisement
  Interventions: Diagnostic Test: Diagnostic Test
- Subjective cognitive decline: Individuals who subjectively experience cognitive decline but do not show deficits in age-, sex- and education-normed neuropsychological test results. Those individuals are part of the DELCODE cohort and were initially recruited in a memory clinic.
  Interventions: Diagnostic Test: Diagnostic Test
- Mild cognitive impairment: Individuals who show deficits in neuropsychological test procedures but who do not exhibit substantial problems in daily life. Those individuals are part of the DELCODE cohort and were initially recruited in a memory clinic.
  Interventions: Diagnostic Test: Diagnostic Test
- Dementia due to Alzheimer's disease: Individuals diagnosed with dementia due to Alzheimer's disease by relying on anamnesis, neuropsychological test results, results of MRI and biomarkers found in the cerebrospinal fluid. Those individuals are part of the DELCODE cohort and were initially recruited in a memory clinic.
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Diagnostic Test: Contrast agentenhanced MRI using Gadovist by using the contrast agent Gadovist we aim to visualize the blood-brain barrier. Furthermore, we aim to measure a newly developed biomarker of the blood-brain barrier in the cerebro-spinal fluid. And sleep quality measurement with a polysomnography.

SUMMARY:
The aim of our study is the analysis of sleep phases and quality as well as the detection of respiratory pauses in subjects with cognitive disorder. To assess whether sleep quality is associated with the blood-brain barrier and Alzheimer's disease, which may be indicative of an early, non-invasively measurable change in brain activity in the early stages of Alzheimer's disease.

DETAILED DESCRIPTION:
The aim of our study is the analysis of sleep phases and quality as well as the detection of respiratory pauses in subjects with cognitive disorder. To assess whether sleep quality is associated with the blood-brain barrier and Alzheimer's disease, which may be indicative of an early, non-invasively measurable change in brain activity in the early stages of Alzheimer's disease.

Sleep quality impairment is a known risk factor for memory impairment. There is increasing evidence of a link between measurable sleep parameters, in particular a reduction of slow waves of deep sleep in cognitive deficits. Also, breathing pauses during sleep are associated with increased daytime sleepiness and cognitive impairment. This observational study is intended to establish a possible link between subjective memory disturbances and altered sleep quality or respiratory breaks during sleep. In the run-up to this study, they performed a special MRI scan of the head and a lumbar puncture (removal of nerve water) in a different context. The aim of this imaging study and the new biomarker in brain water was to investigate the function of the blood-brain barrier that occurs in Alzheimer's disease. The results of the studies on the quality of sleep should be evaluated in the context of this study in connection with the findings of the MRI examination and lumbar puncture.

ELIGIBILITY:
The eligibility criteria are defined by the study protocol from the observational study DZNE - Longitudinal Cognitive Impairment and Dementia Study (DELCODE).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A description of the study population is provided by DZNE - Longitudinal Cognitive Impairment and Dementia Study (DELCODE).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Marker of blood-brain dysfunction using MRI | 1 day
  Dynamic T1 contrast enhanced sequence using Gadovist
Markers of blood-brain dysfunction using CSF | 1 day
  Platelet-derived growth factor receptor-β in CSF
Sleep quality measurement | 2 day
  Polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No